CLINICAL TRIAL: NCT05493189
Title: Assessment of CPR Skills Acquisition and Retention: Impact of Technology and Self-training
Acronym: TrainCPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Rede de Investigação em Saúde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TrainCPR
Record Dates: First submitted 2022-08-01; First posted 2022-08-09 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Cardiopulmonary resuscitation; Chest compressions; Acquisition; Retention

STUDY DESIGN:
Intervention Model Description: Experimental case-control study, aligned in two phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants with no additional autonomous training sessions.
- Intervention Group (Experimental): Participants exposed to 2 additional autonomous training sessions (after 2 and 6 months).
  Interventions: Other: Additional autonomous training sessions

INTERVENTIONS:
Other: Additional autonomous training sessions — The duration of the autonomous training will be 30 minutes, using a feedback CPR training simulator (eg Laerdal Little Anne QCPR).
  Arms: Intervention Group

SUMMARY:
Cardiopulmonary resuscitation (CPR) is an emergency maneuver used on a victim who is in cardiac arrest. Early and efficient CPR, with a focus on chest compressions, is a key element in increasing victim survival. The success of resuscitation does not only depend on the immediate initiation of the maneuvers, but also on the quality with which they are applied. However, there is an obvious gap in the knowledge of these maneuvers. This study aims to analyze the acquisition and retention/maintenance of cardiopulmonary resuscitation (CPR) skills and the impact of the use of technology and autonomous training in medical students.

DETAILED DESCRIPTION:
The objectives of this study include:

1. Study the impact of using technology, namely simulators with automatic feedback, in CPR training.
2. Study the potential of autonomous training as a complementary and/or alternative methodology in CPR training.
3. Assess the acquisition and retention/maintenance of CPR skills, through autonomous and regular training.

The findings of this project are expected to promote awareness and behavioral change in the rescuer, leading to better outcomes for patients.

Experimental case-control study, aligned in two phases. In a first phase, all participants will be exposed to a period of autonomous training, with measurements of performance and quality of CPR, before and after training. This phase will allow investigating the acquisition of skills through autonomous training and leveling the skills of the entire sample. In a second phase, the sample will be randomly distributed between two groups and the retention/maintenance of skills will be evaluated over 1 year, considering that one of the groups will be exposed to 2 additional autonomous training sessions (after 2 and 6 months). The collection of technical skills data will be performed in the pre-training period, post-training (time zero) and after 2, 6 and 12 months - corresponding to 5 data collection moments, in both groups.

Both autonomous training and technical skills data collection will take place using a feedback CPR training simulator (eg Laerdal Little Anne QCPR). Along with the collection of technical skills data, theoretical knowledge will be assessed through a questionnaire. The duration of the autonomous training will be 30 minutes.

The sample will be recruited by convenience (non-probabilistic sample), using students of the 4th year of the Integrated Master in Medicine of the Faculty of Medicine of the University of Porto.

Data collection will take place at the Clinical Simulation Center of the Faculty of Medicine of the University of Porto (Portugal);

An estimate of the sample size was calculated considering the use of an ANOVA test for repeated measures. Using the G-Power software and considering an effect size of 0.20, significance level of 0.05, power of 0.95, for two groups and five measures, 96 participants will be needed. In this calculation, a null correlation coefficient was used, opting for a conservative approach to sample size calculation. Anticipating eventual dropouts, 150 participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>= 18 years of age);
* Good state of health;
* Lack of formal training in CPR.

Exclusion Criteria:

* Pregnant women;
* Individuals with reduced mobility;
* Physical fatigue and/or reported muscle pain;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in CPR skills (acquisition) | Measurements of performance and quality of CPR (2 minutes of continuous chest compressions), immediately before and immediately after training, during the first phase (before randomization and group allocation).
  Technical skills data collection will take place using a feedback CPR training simulator (eg Laerdal Little Anne QCPR). Along with the collection of technical skills data, theoretical knowledge will be assessed through a questionnaire. Both technical skills and theoretical knowledge will be aggregated to one general skills score.
Difference in CPR skills retention | Measurements of performance and quality of CPR (2 minutes of continuous chest compressions), in second phase at 2, 6 and 12 months.
  Technical skills data collection will take place using a feedback CPR training simulator (eg Laerdal Little Anne QCPR). Along with the collection of technical skills data, theoretical knowledge will be assessed through a questionnaire. Both technical skills and theoretical knowledge will be aggregated to one general skills score.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Sa-Couto, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Faculty of Medicine (FMUP), Porto, Portugal

IPD SHARING:
Plan to Share IPD: No